CLINICAL TRIAL: NCT04027309
Title: A Phase 3, Multicenter, Open-label, Randomized, Study of Gilteritinib Versus Midostaurin in Combination With Induction and Consolidation Therapy Followed by One-year Maintenance in Patients With Newly Diagnosed Acute Myeloid Leukemia (AML) or Myelodysplastic Syndromes With Excess Blasts-2 (MDS-EB2) With FLT3 Mutations Eligible for Intensive Chemotherapy (HOVON 156 AML / AMLSG 28-18)
Brief Title: A Study of Gilteritinib Versus Midostaurin in Combination With Induction and Consolidation Therapy Followed by One-year Maintenance in Patients With Newly Diagnosed Acute Myeloid Leukemia or Myelodysplastic Syndromes With Excess Blasts-2 With FLT3 Mutations Eligible for Intensive Chemotherapy
Acronym: HOVON 156 AML
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Stichting Hemato-Oncologie voor Volwassenen Nederland (Other)
Collaborators: Deutsch-Österreichische Studiengruppe Akute Myeloische Leukämie (AMLSG) (Unknown); Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HO156; 2018-000624-33 (EudraCT Number); AMLSG 28-18 (Other: AMLSG); Pasha (Other: Astellas)
Record Dates: First submitted 2019-07-18; First posted 2019-07-19 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-09

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndrome With Excess Blasts-2
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — gilteritinib; midostaurin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (Midostaurin) (Active Comparator): Midostaurin (50 mg BID PO) - Cycle 1 (day 8-21), Cycle 2 (day 8-21), Consolidation (only during chemo consolidation (day 8-21 - with max of 3 cycles), Maintenance (day 1-365)
  Interventions: Drug: Midostaurin
- Arm B (Gilteritinib) (Experimental): Gilteritinib (120 mg QD PO) - Cycle 1 (day 8-21), Cycle 2 (day 8-21), Consolidation (only during chemo consolidation (day 8-21 - with max of 3 cycles), Maintenance (day 1-365)
  Interventions: Drug: Gilteritinib

INTERVENTIONS:
Drug: Gilteritinib — Patients with a FLT3 mutation w ill be randomized to receive either the investigational drug gilteritinib or midostaurin given sequentially to standard induction and consolidation chemotherapy. After completing induction and consolidation treatment, patients who achieve CR/CRi/MLFS will receive maintenance therapy with gilteritinib or midostaurin
  Other Names: ASP2215
  Arms: Arm B (Gilteritinib)
Drug: Midostaurin — Patients with a FLT3 mutation w ill be randomized to receive either the investigational drug gilteritinib or midostaurin given sequentially to standard induction and consolidation chemotherapy. After completing induction and consolidation treatment, patients who achieve CR/CRi/MLFS will receive maintenance therapy with gilteritinib or midostaurin
  Other Names: Rydapt
  Arms: Arm A (Midostaurin)

SUMMARY:
Activating mutations in the fms like tyrosine kinase 3 (FLT3) gene are observed in approximately 30% of patients with newly diagnosed acute myeloid leukemia (AML). Addition of the multitargeted kinase inhibitor midostaurin to standard chemotherapy prolongs event-free survival (EFS) and overall survival (OS) in patients with a FLT3 mutation. Gilteritinib is a more potent and more specific inhibitor of mutant FLT3 in comparison to midostaurin and has shown promising clinical activity in AML.

DETAILED DESCRIPTION:
AML and MDS-EB2 are malignant diseases of the bone marrow. The standard treatment for these diseases is chemotherapy. A subgroup of these diseases is characterized by a specific error in the DNA of the leukemic cells. This is the FLT3 mutation, which leads to a change of a certain protein (FLT3) on the blasts. This altered protein plays an important role in the development of leukemia and the survival of leukemic cells.

FLT3 can be inhibited by the drug midostaurin. Adding midostaurin to chemotherapy leads to better treatment results in patients with AML. Therefore, the standard treatment for AML or MDS-EB2 with a FLT3 mutation (FLT3-AML) is a combination of chemotherapy and midostaurin.

Gilteritinib is also a drug that inhibits FLT3. In laboratory studies, gilteritinib was found to be significantly more specific and potent than midostaurin in inhibiting FLT3.

Gilteritinib has subsequently been studied in patients with AML, who relapsed after previous treatment with chemotherapy. This resulted in a much larger number of complete remissions than previously seen when comparable patients were treated with midostaurin.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Newly diagnosed AML or MDS with excess of blasts-2 (EB2) defined according to WHO criteria (appendix A), with centrally documented FLT3 gene mutation (either TKD or ITD or both). AML may be secondary to prior hematological disorders, including MDS, and/or therapy-related. Patients may have had previous treatment with erythropoiesis stimulating agents (ESA) or hypomethylating agents (HMAs) for an antecedent phase of MDS. ESA and HMAs have to be stopped at least four weeks before registration.
* FLT3 mutation as assessed by DNA fragment analysis PCR for FLT3-ITD and FLT3-TKD mutation. Positivity is defined as a FLT3-ITD or FLT3-TKD / FLT3-WT ratio of ≥ 0.05 (5%).
* Considered to be eligible for intensive chemotherapy
* Patient is suitable for oral administration of study drug
* WHO/ECOG performance status ≤ 2
* Adequate hepatic function as evidenced by

  * Serum total bilirubin ≤ 2.5 × upper limit of normal (ULN) unless considered due to leukemic involvement following written approval by the (co) Principal Investigator
  * Aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase (ALP) ≤ 3.0 × ULN, unless considered due to leukemic involvement following written approval by the (co) Principal Investigator
* Adequate renal function as defined by creatinine clearance > 40 mL/min based on the Cockroft-Gault glomerular filtration rate (GFR)
* Written informed consent
* Patient is capable of giving informed consent
* Female patient must either:

  * Be of nonchildbearing potential:

    * Postmenopausal (defined as at least 1 year without any menses) prior to screening, or
    * Documented surgically sterile or status posthysterectomy (at least 1 month prior to screening)
  * Or, if of childbearing potential,

    * Agree not to try to become pregnant during the study and for 6 months after the final study drug administration
    * And have a negative urine or serum pregnancy test at screening
    * And, if heterosexually active, agree to consistently use highly effective* contraception per locally accepted standards in addition to a barrier method starting at screening and throughout the study period and for 6 months after the final study drug administration.
    * Highly effective forms of birth control include:

      * Consistent and correct usage of established hormonal contraceptives that inhibit ovulation,
      * Established intrauterine device (IUD) or intrauterine system (IUS),
      * Bilateral tubal occlusion,
      * Vasectomy (A vasectomy is a highly effective contraception method provided the absence of sperm has been confirmed. If not, an additional highly effective method of contraception should be used.)
      * Male is sterile due to a bilateral orchiectomy.
      * Sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual activity during the entire period of risk associated with the study drug. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical study and the preferred and usual lifestyle of the patient.
    * (*)List is not all inclusive. Prior to enrollment, the investigator is responsible for confirming patient will utilize highly effective forms of birth control per the requirements of the CTFG Guidance document 'Recommendations related to contraception and pregnancy testing in clinical trials', September 2014 (and any updates thereof) during the protocol defined period.
  * Female patient must agree not to breastfeed starting at screening and throughout the study period, and for 2 months and 1 week after the final study drug administration.
  * Female patient must not donate ova starting at screening and throughout the study period, and for 6 months after the final study drug administration.
* Male patient and their female partners who are of childbearing potential must be using highly effective contraception per locally accepted standards in addition to a barrier method starting at screening and continue throughout the study period and for 4 months and 1 week after the final study drug administration.
* Male patient must not donate sperm starting at screening and throughout the study period and for 4 months and 1 week after the final study drug administration.
* Patient agrees not to participate in another interventional study while on treatment

Exclusion Criteria:

* Prior chemotherapy for AML or MDS-EB2, including prior treatment with hypomethylating agents. Hydroxyurea is allowed for the control of peripheral leukemic blasts in patients with leukocytosis (e.g., white blood cell [WBC] counts > 30 x 10^9/L)
* Acute promyelocytic leukemia (APL) with PML-RARA or one of the other pathognomonic variant fusion genes/chromosome translocations
* Blast crisis after CML
* Known or suspected hypersensitivity to midostaurin or gilteritinib and/or any excipients
* Patient requires treatment with concomitant drugs that are strong inducers of cytochrome P450 (CYP) 3A
* Breast feeding at start of study treatment
* Active infection, including hepatitis B or C or HIV infection that is uncontrolled at randomization. An infection controlled with an approved or closely monitored antibiotic/antiviral/antifungal treatment is allowed.
* Patients with a currently active second malignancy. Patients are not considered to have a currently active malignancy if they have completed therapy and are considered by their physician to be at less than 30% risk of relapse within one year. However, patients with the following history/concurrent conditions are allowed:

  * Basal or squamous cell carcinoma of the skin;
  * Carcinoma in situ of the cervix;
  * Carcinoma in situ of the breast;
  * Incidental histologic finding of prostate cancer
* Significant active cardiac disease within 6 months prior to the start of study treatment, including:

  * New York Heart Association (NYHA) Class III or IV congestive heart failure;
  * Myocardial infarction;
  * Unstable angina and/or stroke;
  * Left ventricular ejection fraction (LVEF) < 40% by ECHO or MUGA scan obtained within 28 days prior to the start of study treatment
* QTc interval using Fridericia's formula (QTcF) ≥ 450 msec (average of triplicate determinations) or other factors that increase the risk of QT prolongation or arrhythmic events (e.g., heart failure, family history of long QT interval syndrome). Prolonged QTc interval associated with bundle branch block or pacemaking is permitted with written approval of the (co) Principal Investigator.
* Patient with hypokalemia and/or hypomagnesemia before registration (defined as values below LLN) Note: electrolyte suppletion is allowed to correct LLN values before registration.
* Dysphagia, short-gut syndrome, gastroparesis, or other conditions that limit the ingestion or gastrointestinal absorption of orally administered drugs
* Clinical symptoms suggestive of active central nervous system (CNS) leukemia or known CNS leukemia. Evaluation of cerebrospinal fluid (CSF) during screening is only required if there is a clinical suspicion of CNS involvement by leukemia during screening
* Immediate life-threatening, severe complications of leukemia such as uncontrolled bleeding and/or disseminated intravascular coagulation
* Any other medical or psychological condition deemed by the Investigator to be likely to interfere with a patient's ability to give informed consent or participate in the study
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 777 (Actual)
Dates: Start 2019-12-20 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2033-06 (Estimated)

PRIMARY OUTCOMES:
Overal survival (OS) | Approximately up to 70 months following first patient enrolment
  Overall survival (OS), defined as the time from date of randomization to the date of death due to any cause. Patients still alive or lost to follow up will be censored at the time they were last known to be alive.

SECONDARY OUTCOMES:
Event-free survival (EFS) | Approximately up to 70 months following first patient enrolment
  Event-free survival (EFS), defined as the time from randomization to failure to achieve CR after remission induction, death or relapse after achieving CR, whichever occurs first. A patient is said to have failed to achieve CR after remission induction if his/her best response during or at completion of the induction therapy is less than CR. Patients who achieved CR after remission induction and are not known to have relapsed or died will be censored at the date of last clinical assessment. CR is determined by the Investigator according to the European LeukemiaNet (ELN2017) recommended response criteria.
CR rate after remission induction | Approximately up to 70 months following first patient enrolment
  CR rate after remission induction is defined as the percentage of patients with best response of CR during or at completion of induction therapy.
EFS with modified CR (mEFS) | Approximately up to 70 months following first patient enrolment
  EFS with modified CR (mEFS) is defined similarly to EFS above. It is the time from randomization to failure to achieve CR after remission induction, death or relapse after achieving CR, whichever occurs first. However, a patient will be considered to have failed to achieve CR after remission induction if CR is not achieved within 60 days after the start of the last induction cycle. Patients who achieve CR within 60 days of the start of the last induction cycle and are not known to have relapsed or died will be censored at the date of last clinical assessment.
CR and CRi rates after induction cycle 1 and after induction cycle 2 | Approximately up to 70 months following first patient enrolment
  CR and CRi are determined by the Investigator based on the European LeukemiaNet (ELN2017) recommended response criteria.
Relapse-free survival (RFS) after CR | Approximately up to 70 months following first patient enrolment
  RFS is defined as time from the date of achievement of CR as determined by the Investigator until relapse or death from any cause, whichever comes first. Patients still in first CR and alive or lost to follow up will be censored at the date of last clinical assessment.
Cumulative incidence of relapse (CIR) after CR | Approximately up to 70 months following first patient enrolment
  CIR is measured from the date of achievement of CR as determined by the Investigator until the date of relapse. Patients not known to have relapsed will be censored on the date of last clinical assessment. Patients who died without relapse will be counted as a competing cause of failure.
Cumulative incidence of death (CID) after CR | Approximately up to 70 months following first patient enrolment
  CID is measured from the date of achievement of CR as determined by the Investigator until the date of death from any cause. Patients not known to have died will be censored on the date they were last known to be alive. Patients who experienced relapse in CR will be counted as competing cause of failure.
CR without minimal residual disease (CRMRD-) rate after induction cycle 2 | Approximately up to 70 months following first patient enrolment
  CRMRD- rate is defined as the percentage of patients who achieved CR as determined by the Investigator with no evidence of MRD
CR or CRi without minimal residual disease (CR/CRiMRD-) rate after induction cycle 2 | Approximately up to 70 months following first patient enrolment
  CR or CRi without minimal residual disease (CR/CRiMRD-) rate after induction cycle 2, defined as the percentage of patients who achieved CR or CRi as determined by the Investigator with no evidence of MRD
Frequency and severity of adverse events according to CTCAE v5.0 | Continuously throughout the study, starting from informed consent until 30 days following the last administration of any study drug
  Adverse events will be evaluated using the National Cancer Institute's Common Terminology Criteria for AEs (CTCAE) version 5.0
Time to hematopoietic recovery after each chemotherapy treatment cycle | Approximately up to 70 months following first patient enrolment
  Time to hematopoietic recovery is defined as the time from the start of the cycle until recovery
Allogeneic stem cell transplantation (allo-SCT) rate | Approximately up to 70 months following first patient enrolment
  Allo-SCT rate is defined as the percentage of patients who underwent an allo-SCT
Individual domain scores and visual analogue scale (VAS) score of the European Quality of Life 5 Dimensions (EQ-5D-5L) Questionnaire | At entry, 1st day of maintenance and every 3 months during maintenance until relapse or treatment discontinuation (approximately up to 70 months following first patient enrolment)
  The EQ-5D-5L is a 5 item questionnaire that assesses 5 domains including mobility, self-care, usual activities, pain/discomfort and anxiety/depression plus a visual analog scale rating "health today". Each domain has 5 levels. Each level has a 1 digit number expressing the level selected for that domain. These levels are summed up and the self-rated health is recorded on a 20 cm vertical, visual analogue scale, with endpoints labelled "the best health you can imagine" and "the worst health you can imagine".
Individual subdomain scores and the global health status/QoL scale of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) | At entry, 1st day of maintenance and every 3 months during maintenance until relapse or treatment discontinuation (approximately up to 70 months following first patient enrolment)
  The EORTC QLQ-C30 is a 30-item questionnaire that assesses 5 functional subdomains (physical functioning, role functioning, emotional functioning, cognitive functioning and social functioning), 1 global health status, 3 symptom subdomains (fatigue, nausea and vomiting and pain) and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). Most of the 30 items have 4 response levels (1="not at all", 2="a little", 3="quite a bit", and 4="very much"), with 2 questions relying on a 7-point numeric rating scale from 1="very poor" to 7="excellent". Raw scores are transformed into scale scores ranging from 0 to 100, with higher scores representing better functioning/QoL or worse symptom burden.

CONTACTS AND LOCATIONS:
Overall Officials: M. Raaijmakers, Prof. Dr., Principal Investigator — Erasmus MC / HOVON
Locations (193):
- Australia (24):
  - AU-Adelaide-FLINDERS, Adelaide
  - AU-Adelaide-RAH, Adelaide
  - AU-Brisbane-PAH, Brisbane
  - AU-Brisbane-RBWH, Brisbane
  - AU-Camperdown-RPA, Camperdown
  - AU-Douglas-TOWNSVILLE, Douglas
  - AU-Geelong VIC-BARWONHEALTH, Geelong
  - AU-Gosford NSW-GOSFORDHOSPITAL, Gosford
  - AU-Hobart TAS-RHOBART, Hobart
  - AU-Melbourne-ALFRED, Melbourne
  - AU-Melbourne-AUSTIN, Melbourne
  - AU-Melbourne-BOXHILL, Melbourne
  - AU-Melbourne-MONASH, Melbourne
  - AU-Melbourne-RMELBOURNE, Melbourne
  - AU-Melbourne-SVHM, Melbourne
  - AU-Perth-FSH, Perth
  - AU-Perth-RPH, Perth
  - AU-Perth-SCGH, Perth
  - AU-Sydney-CONCORD, Sydney
  - AU-Sydney-NEPEAN, Sydney
  - AU-Sydney-RNSH, Sydney
  - AU-Sydney-WSAH, Sydney
  - St George Hospital, Sydney
  - AU-Waratah-CALVARYMATER, Waratah
- Austria (6):
  - AT-Graz-MEDUNIGRAZ, Graz
  - AT-Innsbruck-IMED, Innsbruck
  - AT-Linz-KEPLER, Linz
  - AT-Linz-ORDENSKLINIKUM, Linz
  - AT-Salzburg-SALK, Salzburg
  - AT-Vienna-HANUSCH, Vienna
- Belgium (13):
  - BE-Antwerpen-ZNASTUIVENBERG, Antwerp
  - BE-Brugge-AZBRUGGE, Bruges
  - BE-Brussel-BORDET, Brussels
  - BE-Bruxelles-STLUC, Brussels
  - BE-Gent-UZGENT, Ghent
  - BE-Haine-Saint-Paul-JOLIMONT, Haine-Saint-Paul
  - BE-Hasselt-VIRGAJESSE, Hasselt
  - BE-Leuven-UZLEUVEN, Leuven
  - BE-Liege-CHRCITADELLE, Liège
  - BE-Liege-CHULIEGE, Liège
  - BE-Mons-AMBROISE, Mons
  - BE-Roeselare-AZDELTA, Roeselare
  - BE-Yvoir-MONTGODINNE, Yvoir
- Finland (2):
  - FI-Helsinki-HUS, Helsinki
  - FI-Tampere-TAYS, Tampere
- France (32):
  - FR-Amiens-CHUAMIENS, Amiens
  - FR-Angers-CHUANGERS, Angers
  - FR-Argenteuil-CHARGENTEUIL, Argenteuil
  - FR-Bayonne-CHCOTEBASQUE, Bayonne
  - FR-Besançon Cedex-JEANMINJOZ, Besançon
  - FR-Bobigny-AVICENNE, Bobigny
  - FR-Le Chesnay cedex-CHVERSAILLES, Chesnay
  - FR-Clamart-HIAPERCY, Clamart
  - FR-Clermont-Ferrand-ESTAING, Clermont-Ferrand
  - FR-Grenoble cedex 9-CHUGRENOBLE, Grenoble
  - FR-Lille-CHULILLE, Lille
  - FR-Limoges-CHULIMOGES, Limoges
  - FR-Lyon Pierre Benite cedex-LYONSUD, Lyon
  - FR-Lyon-LEONBERARD, Lyon
  - FR-Marseille-IPC, Marseille
  - FR-Montpellier-STELOI, Montpellier
  - FR-Nantes-CHUNANTES, Nantes
  - FR-Nice-CAL, Nice
  - FR-Nice-LARCHET, Nice
  - FR-Paris cedex 10-SAINTLOUIS, Paris
  - FR-Paris cedex 15-NECKER, Paris
  - FR-Pessac Cedex-CHUBORDEAUX, Pessac
  - FR-Poitiers-CHUPOITERS, Poitiers
  - FR-Reims-CHREIMS, Reims
  - FR-Rennes cedex 9-CHURENNES, Rennes
  - FR-Rouen cedex-BECQUEREL, Rouen
  - FR-Saint-Priest-en-Jarez-ICLOIRE, Saint-Priest-en-Jarez
  - FR-Strasbourg cedex-HAUTEPIERRE, Strasbourg
  - FR-Toulouse-CHUTOULOUSE, Toulouse
  - FR-Tours cedex-BRETONNEAU, Tours
  - FR-Vandoeuvre Les Nancy-CHRUNANCY, Vandœuvre-lès-Nancy
  - FR-Villejuif-GUSTAVEROUSSY, Villejuif
- Germany (54):
  - DE-Aschaffenburg-KLINIKUMAB, Aschaffenburg
  - DE-Bad Saarow-HELIOSBADSAAROW, Bad Saarow
  - DE-Berlin-CAMPUSBENFRANKLIN, Berlin
  - DE-Berlin-CAMPUSMITTE, Berlin
  - DE-Berlin-CAMPUSVIRCHOW, Berlin
  - DE-Berlin-VIVANTESNEUKOLLN, Berlin
  - DE-Berlin-VIVANTESURBAN, Berlin
  - DE-Bochum-RUB, Bochum
  - DE-Bonn-UNIBONN, Bonn
  - DE-Braunschweig-KLINIKUMBRAUNSCHWEIG, Braunschweig
  - DE-Bremen-KBM, Bremen
  - DE-Darmstadt-KLINIKUMDARMSTADT, Darmstadt
  - DE-Dortmund-JOHODORTMUND, Dortmund
  - DE-Düsseldorf-MEDUNIDUESSELDORF, Düsseldorf
  - DE-Essen-KEM, Essen
  - DE-Esslingen-KLINIKUMESSLINGEN, Esslingen am Neckar
  - DE-Flensburg-MALTESER, Flensburg
  - DE-Frankfurt-KLINIKUMFRANKFURT, Frankfurt
  - DE-Giessen-UKGM, Giessen
  - DE-Goch-KKLE, Goch
  - DE-Greifswald-UNIGREIFSWALD, Greifswald
  - DE-Hamburg-ASKLEPIOSSTGEORG, Hamburg
  - DE-Hamburg-ASKLEPIOS, Hamburg
  - DE-Hamburg-UKE, Hamburg
  - DE-Hamm-EVKHAMM, Hamm
  - DE-Hanau-KLINIKUMHANAU, Hanau
  - DE-Hannover-MHHANNOVER, Hanover
  - DE-Hannover-SILOAHKRH, Hanover
  - DE-Heilbronn-SLK, Heilbronn
  - DE-Herne-MARIENHOSPITALHERNE, Herne
  - DE-Homburg-UNIKLINIKSAARLAND, Homburg
  - DE-Kaiserslautern-WESTPFALZ, Kaiserslautern
  - DE-Karlsruhe-KLINIKUMKARLSRUHE, Karlsruhe
  - DE-Lemgo-KLINIKUMLIPPE, Lemgo
  - DE-Ludwigshafen-KLILU, Ludwigshafen
  - DE-Lübeck-UKSHLUBECK, Lübeck
  - DE-Luedenscheid-KLINIKUMLUEDENSCHEID, Lüdenscheid
  - DE-Magdeburg-OVGU, Magdeburg
  - DE-Mainz-UNIMEDIZINMAINZ, Mainz
  - DE-Meschede-HOCHSAUERLAND, Meschede
  - DE-Minden-MUEHLENKREISKLINKEN, Minden
  - DE-München-IRZTUM, München
  - DE-Offenburg-ORTENAUKLINIKUM, Offenburg
  - DE-Oldenburg-KLINIKUMOLDENBURG, Oldenburg
  - DE-Passau-KLINIKUMPASSAU, Passau
  - DE-Regensburg-UKR, Regensburg
  - DE-Saarbrücken-CARITASKLINIKUM, Saarbrücken
  - DE-Stuttgart-DIAKSTUTTGART, Stuttgart
  - DE-Stuttgart-KLINIKUMSTUTTGART, Stuttgart
  - DE-Trier-MUTTERHAUS, Trier
  - DE-Tübingen-MEDUNITUEBINGEN, Tübingen
  - DE-Ulm-UNIKLINKULM, Ulm
  - DE-Villingen-Schwenningen-SBKVS, Villingen-Schwenningen
  - DE-Wuppertal-HELIOSGESUNDHEIT, Wuppertal
- Ireland (8):
  - IE-Cork-CUH, Cork
  - IE-Dublin 24-TUH, Dublin
  - IE-Dublin 4-SVUH, Dublin
  - IE-Dublin 7-MATER, Dublin
  - IE-Dublin 8-STJAMES, Dublin
  - IE-Dublin 9-BEAUMONT, Dublin
  - IE-Galway-UHGALWAY, Galway
  - IE-Co. Limerick-UHL, Limerick
- LT-Vilnius-SANTA, Vilnius, Lithuania
- Netherlands (21):
  - NL-Den Bosch-JBZ, 's-Hertogenbosch
  - NL-Amersfoort-MEANDERMC, Amersfoort
  - NL-Amsterdam-AMC, Amsterdam
  - NL-Amsterdam-OLVG, Amsterdam
  - NL-Amsterdam-VUMC, Amsterdam
  - NL-Arnhem-RIJNSTATE, Arnhem
  - NL-Breda-AMPHIA, Breda
  - NL-Delft-RDGG, Delft
  - NL-Dordrecht-ASZ, Dordrecht
  - NL-Eindhoven-MAXIMAMC, Eindhoven
  - NL-Enschede-MST, Enschede
  - NL-Groningen-UMCG, Groningen
  - NL-Leeuwarden-MCL, Leeuwarden
  - NL-Leiden-LUMC, Leiden
  - NL-Maastricht-MUMC, Maastricht
  - NL-Nieuwegein-ANTONIUS, Nieuwegein
  - NL-Nijmegen-RADBOUDUMC, Nijmegen
  - NL-Rotterdam-ERASMUSMC, Rotterdam
  - NL-Den Haag-HAGA, The Hague
  - NL-Utrecht-UMCUTRECHT, Utrecht
  - NL-Zwolle-ISALA, Zwolle
- Norway (5):
  - NO-Bergen-HELSEBERGEN, Bergen
  - NO-Oslo-OSLOUH, Oslo
  - NO-Stavanger-HELSESTAVANGER, Stavanger
  - NO-Tromsø-NORTHNOORWEGEN, Tromsø
  - NO-Trondheim-STOLAV, Trondheim
- Spain (14):
  - ES-Barcelona-CLINICUB, Barcelona
  - ES-Barcelona-GERMANTRIALS, Barcelona
  - ES-Barcelona-ICODURANREYNALS, Barcelona
  - ES-Barcelona-MUTUATERRASSA, Barcelona
  - ES-Barcelona-PARCDESALUTMAR, Barcelona
  - ES-Barcelona-SANTPAU, Barcelona
  - ES-Barcelona-VHEBRON, Barcelona
  - ES-Girona-ICSTRUETA, Girona
  - ES-Lleida-ICSVILANOVA, Lleida
  - ES-Madrid-CSGREGORIOMARANON, Madrid
  - ES-Palma-HSLL, Palma
  - ES-Palma-SSIB, Palma
  - ES-Tarragona-JOAN, Tarragona
  - ES-Valencia-MALVARROSA, Valencia
- Sweden (3):
  - SE-Lund-SUH, Lund
  - SE-Stockholm-KAROLINSKAHUDDINGE, Stockholm
  - SE-Uppsala-UPPSALAUH, Uppsala
- Switzerland (10):
  - CH-Aarau-KSA, Aarau
  - CH-Basel-USB, Basel
  - CH-Bellinzona-IOSI, Bellinzona
  - CH-Bern-INSEL, Bern
  - CH-Fribourg-HFR, Fribourg
  - CH-Geneve (14)-HCUGE, Geneva
  - CH-Lausanne-CHUV, Lausanne
  - CH-Luzern-LUKS, Lucerne
  - CH-St. Gallen-KSSG, Sankt Gallen
  - CH-Zürich-USZ, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: HOVON trial website — http://www.hovon.nl